CLINICAL TRIAL: NCT04454671
Title: Efficacy of Ultrasound-guided Percutaneous Neuromodulation Versus Ultrasound-guided Dry Needling of the Suprascapular Nerve in Shoulder Pain
Brief Title: Ultrasound-guided Percutaneous Neuromodulation Versus Dry Needling in Shoulder Pain Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Clinical professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIM/HU/2019/26)
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Shoulder Pain
Keywords: Electric Stimulation Therapy; Dry Needling
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound-guided percutaneous neuromodulation (Experimental): Technique based on electrical stimulation of a peripheral nerve through an ultrasound-guided needle or a muscle at a motor point. The stimulation is performed with low or medium frequency currents in which a sensory and / or motor response is sought by stimulating the peripheral nerve
  Interventions: Other: Ultrasound-guided percutaneous neuromodulation (NMPE)
- Ultrasound-guided dry needling (Placebo Comparator): Dry needling technique applied by ultrasound-guided but without electrical stimulation of a peripheral nerve.
  Interventions: Other: Ultrasound-guided dry needling

INTERVENTIONS:
Other: Ultrasound-guided percutaneous neuromodulation (NMPE) — It is a technique based on electrical stimulation of a peripheral nerve through an ultrasound-guided needle or a muscle at a motor site. The stimulation is performed with low or medium frequency currents in which a sensory and / or motor response is sought by stimulating the peripheral nerve
  Arms: ultrasound-guided percutaneous neuromodulation
Other: Ultrasound-guided dry needling — Dry needling technique under ultrasound imaging in order to ensure accurate placement of the needle for optimum results.
  Arms: Ultrasound-guided dry needling

SUMMARY:
Background: nonspecific shoulder pain is very common and the symptoms can persist for 6 to 12 months in half of patients. Ultrasound-guided Percutaneous Neuromodulation (US-guided PNM) is an intervention based in an electrical stimulation of a peripheral nerve through a needle located close to the target nerve by the use of an ultrasound guidance.

Objectives: the primary aim is to determine changes in strength after US-guided PNM or Ultrasound-guided Dry Needling (US-guided DN) intervention in the Suprascapular Nerve (SN) as well as its effectiveness in changes of muscle function, pain and disability.

Methods: randomised clinical trial (ratio 1:1), single-blind (examiners), parallel, with assessment of third parties. 62 adult participants with unilateral mechanical chronic nonspecific shoulder pain with at least 3-month evolution and shoulder muscle weakness will randomised to one of two procedures: US-guided PNM or US-guided DN. It will be assessed muscle strength, muscle function, pain and disability before, just after, a week and a month after the intervention.

DETAILED DESCRIPTION:
Shoulder pain is the third reason for medical consultation in the world. Many treatment techniques have been proposed. Neuromodulation techniques through the application of an analgesic electric current using a needle as an electrode, are increasingly used in the treatment of pain.

In this study, the investigators will compare whether the application of a neuromodulation technique is more effective than applying the dry needling technique in isolation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic mechanical unilateral shoulder pain of non-specific origin of at least 3 months of evolution
* Weakness in the abduction force and / or external rotation of the shoulder.

Exclusion Criteria:

* Previous shoulder surgery.
* Previous history of shoulder dislocation
* Whiplash.
* Cervical radiculopathy.
* Total rupture of the rotator cuff.
* Adhesive capsulitis.
* Fibromyalgia diagnosis.
* Diabetes.
* Needle phobia or some contraindication for dry needling (anticoagulants or psychiatric disorders).
* Bilateral shoulder pain.
* Pregnancy or having received a dry puncture in the shoulder region in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Muscle Force | Change from Baseline force at 6 month
  Force will be measured by a manual dynamometer (microFET®2, Hoggan Scientific LLC). Measurements will be taken in Newtons (N). It will be evaluated in the movements of external rotation and abduction of both shoulders.
  Manual dynamometry has proven to be a tool with excellent intra-examiner reliability to assess isometric force in external rotation of the shoulder, with an intraclass correlation coefficient (ICC) of 0.96 (0.93-0.98). The minimum value is 0 and de Maximum values is 55

SECONDARY OUTCOMES:
Shoulder Pain | Change from Baseline pain at 6 month.
  Pain intensity will be measured using the Visual Analog Scale (VAS) for pain. The VAS is a 100-mm line, oriented horizontally, with one end representing "no pain" and ten the other end representing "worst pain." Subjects will be asked to rate their current pain with a mark on the scale.
Disability | Change from Baseline disability at 6 month.
  Disability will be measured by Shoulder Pain and Disability Index (SPADI).The Spanish version of SPADI has high test-retest reliability (ICC 0.89-0.93).The clinically important minimum difference varies between 8 and 13.2. The minimum value is 0 and de maximum value is 100
Muscle function | Change from Baseline muscle function at 6 month.
  Muscle function will be measured by an ultrasound scanner (VINNO® E35; VINNO ULTRASOUND S.L.U. ©, Barcelona, Spain) with a linear transducer with a frequency range of 6-16MHz (X6-16L, 5cm footprint) will be used. The unit of measurement used will be millimeters. Muscle thickness at rest and contraction will be measured. On the other hand, the percentage of change in thickness will be measured using the equation (Shrinkage thickness - Rest thickness) * 100 / Rest thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Gallego-Izquierdo, PhD, Study Chair — Alcala University
Locations (2):
- Spain (2):
  - Institut Physiotherapy AND pain, Alcalá de Henares, Madrid
  - Overall Study Officials, Alcalá de Henares, Madrid